CLINICAL TRIAL: NCT05949060
Title: Dating and Sexual Violence Among Sexual Minority Women Living in Central New York (Project DAWN), Study B: Pilot RCT
Brief Title: Effects of Self-Compassion Practice on Stress Reactivity Among Sexual Minority Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: GLMA: Health Professionals Advancing LGBTQ+ Equality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-342 Study B
Record Dates: First submitted 2023-05-23; First posted 2023-07-17 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-11

CONDITIONS: Stress Reaction; Sexuality; Compassion
Keywords: compassion; stress reactivity; sexual minority; gender minority
MeSH Terms: conditions — Fractures, Stress; Sexuality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compassion Intervention (Experimental)
  Interventions: Behavioral: Compassion Intervention
- No Training (No Intervention)

INTERVENTIONS:
Behavioral: Compassion Intervention — The compassion intervention is a single-session 40-min intervention in which the participants practiced soothing rhythm breathing (i.e., they are directed to slow their breathing using a five-count inhale and five-count exhale). They will then be provided didactic instruction on compassion, and will then be guided through an experiential compassion practice adapted that encompasses cultivating feelings of compassion for a loved one and then for oneself.
  Arms: Compassion Intervention

SUMMARY:
This project will test the ability of brief self-compassion training to attenuate physiological and subjective responses to induced stress among sexual minority women, transgender people, and nonbinary people.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Be fluent in English (i.e., speak and read English)
* Have Internet access
* Have a working email address
* Self-identify sexual identity as LGBQ+ or another non-heterosexual identity AND gender identity as cisgender woman, transgender, nonbinary, or other gender minority identity
* Currently live in Central NY

Exclusion Criteria:

* Failing an inclusion criterion
* Report having been hospitalized at an inpatient facility for psychiatric support within the past 6 months
* Report being currently pregnant
* Report a history of heart attack, unstable angina pectoris, heart failure, coronary heart disease, vascular, heart problems, stroke, or brain hemorrhage
* Report being on blood pressure medication
* Have resting systolic blood pressure greater than or equal to 140 mmHg or diastolic blood pressure greater than or equal to 100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who identify as cisgender sexual minority women, transgender, or nonbinary people will be eligible.
Enrollment: 39 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure | Baseline, Immediate Follow-Up (40 minutes after Baseline), During TSST (45-50 minutes after Baseline), Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Systolic and diastolic blood pressure will be measured with an Omron ocillometric blood pressure monitoring device before and after the intervention and before during and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt.
Change in Salivary Cortisol | Baseline, Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Salivary cortisol levels will be collected using Salimetrics saliva swabs before the intervention and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt.
Change in Heart Rate Variability | Baseline, Immediate Follow-Up (40 minutes after Baseline), During TSST (45-50 minutes after Baseline), Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Heart rate variability will be measured with BIOPAC MP160 System before and after the intervention and before during and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt.
Change in Heart Rate | Baseline, Immediate Follow-Up (40 minutes after Baseline), During TSST (45-50 minutes after Baseline), Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Heart rate will be measured with BIOPAC MP160 System before and after the intervention and before during and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt.
Change in Skin Conductance | Baseline, Immediate Follow-Up (40 minutes after Baseline), During TSST (45-50 minutes after Baseline), Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Skin conductance reactivity will be measured with the BIOPAC MP160 System before and after the intervention and before during and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt.
Change in Subjective Stress | Baseline, Immediate Follow-Up (40 minutes after Baseline), Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Subjective stress reactivity will be measured with the six item State-Trait Anxiety Inventory (Marteau & Bekker, 1993), the Positive and Negative Affect Schedule (PANAS), and three visual analog scales before and after the intervention and before during and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt.

SECONDARY OUTCOMES:
Change in PTSD Symptoms | Baseline, Follow-Up (1-month)
  PTSD symptoms will be measured using the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5; Foa et al., 2015). Possible scores on the PDS-5 range from 0 to 80. Higher scores indicate more PTSD symptoms.
Change in Substance Use | Baseline, Follow-Up (1-month)
  Past 30-day substance use, including number of days of any alcohol use, hazardous drinking, cannabis use, prescription drug use, cigarette use, and other drug use was measured using questions from the 2020 National Survey on Drug Use and Health.
Change in Dissociation | Baseline, Immediate Follow-Up (40 minutes after Baseline), Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Change in dissociation will be measured with the five items adapted from scales which measure state dissociation in experience sampling studies (Mason et al., 2017; Vine et al., 2020). Dissociation will be measured before and after the intervention and before and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt. Possible scores for this measure range from 0 to 15. Higher scores indicate more dissociation.
Change in Craving | Baseline, Immediate Follow-Up (40 minutes after Baseline), Immediate Post-TSST (20-30 minutes post-TSST onset), Recovery Post-TSST (10-20 minutes after Immediate Post-TSST time point)
  Change in craving be measured with the 12-item Alcohol Craving Questionnaire - short form - revised (Singleton et al., 1994). Craving will be measured before and after the intervention and before and after participants undergo the Trier Social Stress Test (TSST) modified with a minority stress prompt. Possible scores on this measure range from 12 to 84. Higher scores indicate more alcohol craving.

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Helminen EC, Behari K, Scheer JR. A compassion microintervention targeting stress reactivity among sexual minority women and transgender/nonbinary people: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2024 Oct;145:107660. doi: 10.1016/j.cct.2024.107660. Epub 2024 Aug 8. PMID 39121992